CLINICAL TRIAL: NCT03373149
Title: Growth Hormone Co-treatment Within a GnRH Antagonist Protocol in Patients With Poor Ovarian Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Fertility and Reproductive Health center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gh/poor responders
Record Dates: First submitted 2017-12-07; First posted 2017-12-14 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Infertility, Female
Keywords: IVF; Growth hormone; Poor responders
MeSH Terms: conditions — Infertility, Female | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth hormone/HPuFSH/GnRH antagonist (Experimental): The patients receive growth hormone
  Interventions: Drug: Growth hormone/HPuFSH/GnRH antagonist
- HPuFSH/GnRH antagonist (Active Comparator): Growth hormone is not used
  Interventions: Drug: HPuFSH/GnRH antagonist

INTERVENTIONS:
Drug: Growth hormone/HPuFSH/GnRH antagonist — Growth hormone (Somatropin, Sedico, Egypt) [4 IU/day] and highly purified urinary FSH (HPuFSH) (Fostimon,IBSA, Switzerland) [300 IU/day] will be started on cycle day 3 and will be continued until and including the day of human chorionic gonadotropin (HCG) administration. Starting from cycle day 8, the dose of HPuFSH will be adjusted individually according to ovarian response which will be monitored using transvaginal ultrasound and serum estradiol (E2).
  GnRH antagonist (Cetrorelix acetate) (Cetrotide; Serono International S.A., Geneva, Switzerland) 0.25 mg S.C. once daily will be started when the leading follicle is 14 mm in mean diameter and will be continued until and including the day of HCG administration.
  Arms: Growth hormone/HPuFSH/GnRH antagonist
Drug: HPuFSH/GnRH antagonist — Highly purified urinary FSH (HPuFSH) (Fostimon,IBSA, Switzerland) [300 IU/day] will be started on cycle day 3 and will be continued until and including the day of human chorionic gonadotropin (HCG) administration. Starting from cycle day 8, the dose of HPuFSH will be adjusted individually according to ovarian response which will be monitored using transvaginal ultrasound and serum estradiol (E2).
  GnRH antagonist (Cetrorelix acetate) (Cetrotide; Serono International S.A., Geneva, Switzerland) 0.25 mg S.C. once daily will be started when the leading follicle is 14 mm in mean diameter and will be continued until and including the day of HCG administration.
  Arms: HPuFSH/GnRH antagonist

SUMMARY:
In this study, the investigators will assess the efficacy of growth hormone co-stimulation to GnRH antagonist regimen in poor responders to COH for IVF.

DETAILED DESCRIPTION:
To date, a limited number of studies have been performed in order to assess whether the addition of GH can improve the probability of pregnancy in poor responders undergoing ovarian stimulation for IVF. Moreover, the existing studies are underpowered and, thus, inconclusive.

In this study, the investigators will assess the efficacy of growth hormone co-stimulation to GnRH antagonist regimen in poor responders to COH for IVF.

ELIGIBILITY:
Inclusion Criteria:

* Serum anti-Müllerian hormone (AMH) less than 1.2 ng/ml

Exclusion Criteria:

-

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 228 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
The number of participants who achieved a clinical pregnancy in a transfer cycle | Five weeks after embryo transfer

SECONDARY OUTCOMES:
The number of participants who achieved a ongoing pregnancy in a transfer cycle | Eighteen weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Hisham S Elshaer, Prof., Study Chair — Prof. of Obstetrics and Gynecology,Faculty of medicine, Cairo university. Director of Riyadh Fertility and Reproductive Health center; Usama M Fouda, Prof., Study Director — Prof. of Obstetrics and Gynecology,Faculty of medicine, Cairo university. Consultant at Riyadh Fertility and Reproductive Health center; Mohammad Taymour, M.D, PhD, Principal Investigator — Lecturer of Obstetrics and Gynecology, Faculty of medicine,Cairo university. Consultant at Riyadh Fertility and Reproductive Health center; Ahmed A Wali, M.D, PhD, Principal Investigator — Lecturer of Obstetrics and Gynecology,Faculty of medicine, Cairo university. Consultant at Riyadh Fertility and Reproductive Health center; Fatma Faisel, M.D, PhD, Principal Investigator — Lecturer of Obstetrics and Gynecology,Faculty of medicine, Cairo university. Consultant at Riyadh Fertility and Reproductive Health center
Locations (1):
- Riyadh Fertility and Reproductive Health center, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eftekhar M, Aflatoonian A, Mohammadian F, Eftekhar T. Adjuvant growth hormone therapy in antagonist protocol in poor responders undergoing assisted reproductive technology. Arch Gynecol Obstet. 2013 May;287(5):1017-21. doi: 10.1007/s00404-012-2655-1. Epub 2012 Dec 4. PMID 23208461
- [Derived] Sood A, Mohiyiddeen G, Ahmad G, Fitzgerald C, Watson A, Mohiyiddeen L. Growth hormone for in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD000099. doi: 10.1002/14651858.CD000099.pub4. PMID 34808697